CLINICAL TRIAL: NCT01099254
Title: Effect of Position on Cross Sectional Area of IJV
Brief Title: Internal Jugular Vein Cross Sectional Area
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Gregory A. Schmidt, MD, Roy J. & Lucille A. Carver College of Medicine, University of Iowa
Other Study IDs: 20076778
Record Dates: First submitted 2010-03-29; First posted 2010-04-06 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Central Venous Pressure
Keywords: CVP; US; Trendelenburg position; Ultrasound; Head Down Tilt

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Trendelenburg position is used to distend the central veins, improving both success and safety of vascular cannulation. The purpose of this study is to measure the cross-sectional area of the internal jugular vein (IJV) in three different positions, using surface ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* adult medical or surgical ICU patients who have preexisting central venous (jugular/subclavian only) catheters.

Exclusion Criteria:

* subjects with only a femoral venous catheter.
* subjects whose CVP measurement by the indwelling catheter exceeds 20cm of water.
* subjects younger than 18 years old.
* inability to obtain informed consent from the subject or the subjects authorized representative.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Effect of trendelenburg and reverse trendelenburg position on the cross sectional area of the internal jugular vein | At time of data collection: physiologic study
  There will be substantial anatomic variation in venous size. Further, Trendelenburg positioning will have little impact on venous cross-sectional area in most subjects when compared with supine.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Schmidt, mD, Principal Investigator — Roy J. & Lucille A. Carver College of Medicine, University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Bazaral M, Harlan S. Ultrasonographic anatomy of the internal jugular vein relevant to percutaneous cannulation. Crit Care Med. 1981 Apr;9(4):307-10. doi: 10.1097/00003246-198104000-00004. PMID 7214938
- [Background] Vinayak AG, Levitt J, Gehlbach B, Pohlman AS, Hall JB, Kress JP. Usefulness of the external jugular vein examination in detecting abnormal central venous pressure in critically ill patients. Arch Intern Med. 2006 Oct 23;166(19):2132-7. doi: 10.1001/archinte.166.19.2132. PMID 17060544
- [Derived] Nassar B, Deol GRS, Ashby A, Collett N, Schmidt GA. Trendelenburg position does not increase cross-sectional area of the internal jugular vein predictably. Chest. 2013 Jul;144(1):177-182. doi: 10.1378/chest.11-2462. PMID 23392444